CLINICAL TRIAL: NCT03555838
Title: Improving Hand Function in Chronic SCI With Combined Robotic Training and tDCS
Brief Title: Combined Robotic Training and tDCS in Chronic SCI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Burke Medical Research Institute (Other)
Collaborators: New York State Spinal Cord Injury Research Board (SCIRB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRC549
Record Dates: First submitted 2018-05-15; First posted 2018-06-14 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injuries; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Within-subjects repeated measures design up to 40 SCI participants will be randomized to receive 6-week hand robotic training preceded by 20 min anodal 2mA tDCS or sham (3 sessions/week, 18 sessions total). Randomization will be done using a randomized block design with a block size of 2.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants, raters, and experimenters will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): Participants in this arm will receive 20 minutes of 2 mA transcranial direct current stimulation over the primary motor cortex of the more affected arm prior to robotic training.
  Interventions: Other: transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Participants in this arm will receive 20 minutes of sham transcranial direct current stimulation over the primary motor cortex of the more affected arm prior to robotic training.
  Interventions: Other: sham transcranial direct current stimulation

INTERVENTIONS:
Other: transcranial direct current stimulation — Transcranial direct current stimulation, a form of neuromodulation that uses a low direct current delivered via sponge electrodes on the head.
  Arms: Active tDCS
Other: sham transcranial direct current stimulation — an inactive or placebo version of transcranial direct current stimulation placed on the head via sponge electrodes.
  Arms: Sham tDCS

SUMMARY:
The purpose of this study is to establish the value of combined non-invasive stimulation (tDCS) and behavioral training (robotics) in SCI rehabilitation, and understand the mechanisms of this interaction and its relationship to functional outcome. The investigators hypothesize that supplementary tDCS will augment the functional improvement from robot-training, in chronic SCI.

DETAILED DESCRIPTION:
Study design: Using a within-subjects repeated measures design, up to 40 SCI participants will be randomized to receive 6-week hand robotic training preceded by 20 min anodal 2mA tDCS or sham (3 sessions/week, 18 sessions total). Clinical and functional scales, robotic kinematics and neurophysiological data (TMS evaluation) will be collected before and after the combined intervention period, and a month later (pre, post and follow up evaluations). Randomization will be done using a randomized block design with a block size of 2. All participants, raters, and experimenters will be blinded to treatment allocation.

AIM 1. To determine whether combining non-invasive brain stimulation (tDCS) and behavioral training (robotics) in SCI can lead to functional improvement. The investigators hypothesize that the group receiving the real stimulation will obtain a greater clinical improvement in hand motor function. Using a within subjects repeated measures design, baseline clinical hand function (Box and Blocks test) will be compared to post 6-week robotic training intervention, and then a month later (follow up), each session preceded by real (2mA anodal M1) or sham tDCS.

AIM 2. To examine the kinematic changes (from robotic measures) associated with the combined training. Quantitative measurements obtained from robotics are highly sensitive, precise and reliable. The investigators predict an enhancement of motor performance in all participants, measured by 5 key parameters: mean speed, peak speed, smoothness, aim and deviation; with greater improvements in the intervention group receiving the pre-conditioning effect of transcranial stimulation. These data will identify features of motor control that underlie improvements in clinical function, when comparing the two intervention groups.

AIM 3. To identify and compare the neurophysiological mechanisms (by TMS) associated with the combined training. The relationship between clinical improvement in neurophysiological measures pertaining to robotic motor training alone and combined with tDCS will be assessed. Measuring changes in MEP amplitude of hand muscles before and after the training will establish a) the plasticity associated with training alone and with supplementary brain stimulation, b) the neurophysiological characteristics of patients who respond better to the training. By understanding how brain excitability changes underpin motor dysfunction, and motor recovery, interventions can be more effectively prescribed and prognoses established.

ELIGIBILITY:
Inclusion Criteria:

* Tetraplegia (cervical lesion) with some degree of motor dysfunction in the hand (ability to pick up at least 1 block on the Box and Blocks Test)
* Motor incomplete lesion (measured by the ASIA Impairment Scale, B, C, D)
* Chronic lesion (>6 months after the injury)

Exclusion Criteria:

* Motor and sensory complete lesion (AIS A)
* Presence of potential risk factor for brain stimulation (TMS and tDCS): history of seizures, presence of surgically implanted foreign bodies such as a pacemaker, metal plate in the skull, and metal inside the skull
* History of head trauma and/or cognitive deficit
* Medically unstable

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Box and Blocks Test | Baseline, immediately post-intervention, and 1 month follow up
  A timed functional test to determine gross manual dexterity

SECONDARY OUTCOMES:
Upper Extremity Motor Score | Baseline, immediately post-intervention, and 1 month follow up
  Manual muscle test of arm muscles; Score range from 0= no movement to 5= normal movement.
Spinal Cord Independence Measure (SCIM III) | Baseline, immediately post-intervention, and 1 month follow up
  Evaluates patient's ability to complete activities of daily living; 19 questions in 3 domains; Scored 0 (severely impaired) -100 (independent)
Modified Ashworth Scale | Baseline, immediately post-intervention, and 1 month follow up
  Measures spasticity; Each muscle assessed is scored between 0-4, with 4 indicating rigid limbs or very severely affected.
Nine Hole Peg Test | Baseline, immediately post-intervention, and 1 month follow up
  Timed measure of fine motor skills and dexterity
Questionnaire of von Korff et al Grading the Severity of Chronic Pain | Baseline, immediately post-intervention, and 1 month follow up
  Self-evaluation of pain; 7 questions in total; 0= no pain, 100= severe pain
Quadraplegia Index of Function- Short Form | Baseline, immediately post-intervention, and 1 month follow up
  Global function scale; 6 items dcored on a 5 point scale from 0 (dependent) to 4 (independent).

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to make individual participant data available to other researchers at this time.